CLINICAL TRIAL: NCT01263015
Title: A Randomized, Double-Blind Study of the Safety and Efficacy of GSK1349572 Plus Abacavir/Lamivudine Fixed-Dose Combination Therapy Administered Once Daily Compared to Atripla Over 96 Weeks in HIV-1 Infected Antiretroviral Therapy Naive Adult Subjects
Brief Title: A Trial Comparing GSK1349572 50mg Plus Abacavir/Lamivudine Once Daily to Atripla (Also Called The SINGLE Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114467
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: GSK1349572; Abacavir/Lamivudine; Treatment-naive; HIV Infection; Dolutegravir; integrase inhibitor; Atripla
MeSH Terms: conditions — Infections; HIV Infections | interventions — dolutegravir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination; abacavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dolutegravir (N=~394): (Experimental): Dolutegravir 50mg once daily + abacavir/lamivudine as the fixed-dose combination once daily + Atripla placebo once daily
  Interventions: Drug: Dolutegravir; Drug: Abacavir/Lamivudine; Drug: Atripla placebo
- Atripla (N=~394): (Active Comparator): Atripla once daily + Dolutegravir placebo once daily + abacavir/lamivudine as the fixed-dose combination placebo once daily
  Interventions: Drug: Atripla; Drug: Abacavir/Lamivudine Placebo; Drug: Dolutegravir placebo

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir (also known as GSK1349572) 50 mg taken once daily
  Arms: Dolutegravir (N=~394):
Drug: Atripla — Atripla once daily on an empty stomach
  Arms: Atripla (N=~394):
Drug: Abacavir/Lamivudine — taken once daily; also known as EPZICOM
  Arms: Dolutegravir (N=~394):
Drug: Abacavir/Lamivudine Placebo — matching placebo taken once daily
  Arms: Atripla (N=~394):
Drug: Dolutegravir placebo — matching placebo taken once daily
  Arms: Atripla (N=~394):
Drug: Atripla placebo — matching placebo taken once daily on an empty stomach
  Arms: Dolutegravir (N=~394):

SUMMARY:
The purpose of this trial is to assess the non-inferior antiviral activity of GSK1349572 50 mg plus Abacavir/Lamivudine once daily versus Efavirenz/Emtricitabine/Tenofovir disoproxil fumarate (ATRIPLA® a trade mark of Bristol-Myers Squibb and Gilead Sciences LLC) over 48 weeks; non-inferiority will also be tested at Week 96. This study will be conducted in HIV-1 infected ART-naïve adult subjects. Long term antiviral activity, tolerability, safety, and development of viral resistance will be evaluated.

DETAILED DESCRIPTION:
ING114467 is a Phase 3 randomized, double-blind, double dummy, active-controlled, multicenter, study conducted in approximately 788 HIV-1 infected ART-naïve subjects. Subjects will be randomized 1:1 one of the following treatment arms:

GSK1349572 50 mg plus abacavir/lamivudine fixed-dose combination once daily (approximately 394 subjects)

OR

Atripla once daily (approximately 394 subjects)

Analyses will be conducted at 48 weeks and 96 weeks. Subjects randomized to receive GSK1349572 and who successfully complete 96 weeks of treatment will continue to have access to GSK1349572 plus abacavir/lamivudine fixed-dose combination through the study until it is locally available-as long as they continue to derive clinical benefit, until they meet a protocol-defined reason for discontinuation, or until development of the compound is terminated.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Screening plasma HIV-1 RNA ≥1000 c/mL
* Antiretroviral-naïve (≤ 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection)
* Ability to understand and sign a written informed consent form
* Willingness to use approved methods of contraception to avoid pregnancy (women of child bearing potential only)
* Age equal to or greater than 18 years
* A negative HLAB*5701 allele assessment

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Active Center for Disease and Prevention Control (CDC) Category C disease
* Hepatic impairment
* HBV co-infection
* Anticipated need for HCV therapy during the study
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Malignancy within the past 5 years
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents or any immunomodulator within 28 days of Screening
* Exposure to an agent with documented activity against HIV-1 in vitro or an experimental vaccine or drug within 28 days of first dose of study medication
* Primary viral resistance in the Screening result
* Verified Grade 4 laboratory abnormality
* ALT >5 xULN
* ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin);
* Estimated creatinine clearance <50 mL/min
* Recent history (≤3 months) of upper or lower gastrointestinal bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2011-02-01; Primary Completion 2012-05-14 (Actual); Study Completion 2015-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (114):
- United States (45):
  - GSK Investigational Site, Hobson City, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (4):
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Fitzroy North, Victoria
  - GSK Investigational Site, Prahran, Victoria
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Denmark (3):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense
- France (6):
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tourcoing
- Germany (8):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (6):
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
- Netherlands (2):
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Spain (23):
  - GSK Investigational Site, Oviedo, Principality of Asturias
  - GSK Investigational Site, (Móstoles) Madrid
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Granollers (Barcelona)
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo ( Pontevedra)
- United Kingdom (5):
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Tooting, London

REFERENCES:
- [Background] Brinson C, Walmsley S, Arasteh K, et al. Dolutegravir treatment response and safety by key subgroups in treatment naive HIV-infected individuals. Published at: Conference on Retroviruses and Opportunistic Infections - 20th Annual; March 3-6, 2013; Atlanta, GA.
- [Derived] Walmsley S, Baumgarten A, Berenguer J, Felizarta F, Florence E, Khuong-Josses MA, Kilby JM, Lutz T, Podzamczer D, Portilla J, Roth N, Wong D, Granier C, Wynne B, Pappa K. Brief Report: Dolutegravir Plus Abacavir/Lamivudine for the Treatment of HIV-1 Infection in Antiretroviral Therapy-Naive Patients: Week 96 and Week 144 Results From the SINGLE Randomized Clinical Trial. J Acquir Immune Defic Syndr. 2015 Dec 15;70(5):515-9. doi: 10.1097/QAI.0000000000000790. PMID 26262777
- [Derived] Walmsley SL, Antela A, Clumeck N, Duiculescu D, Eberhard A, Gutierrez F, Hocqueloux L, Maggiolo F, Sandkovsky U, Granier C, Pappa K, Wynne B, Min S, Nichols G; SINGLE Investigators. Dolutegravir plus abacavir-lamivudine for the treatment of HIV-1 infection. N Engl J Med. 2013 Nov 7;369(19):1807-18. doi: 10.1056/NEJMoa1215541. PMID 24195548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consisted of 96 weeks double-blind phase, followed by a 48 week open-label phase.
Pre-assignment Details: A total of 844 participants (par.) were randomized (1:1) to one of the two treatment arms. Of these, 833 par. received at least one dose of study medication. Of the 11 par. who were randomized but not treated with investigational product, 7 par. withdrew consent, 3 par. were randomized in error, and 1 par. was lost to follow-up.
Groups:
- DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily: During double-blind phase, participants received a dolutegravir (DTG) 50 milligram (mg) tablet along with an Abacavir/Lamivudine (ABC/3TC) 600/300 mg tablet once daily (OD) orally, with placebo to match Efavirenz/Tenofovir disoproxil fumarate/Emtricitabine (EFV/TDF/FTC) 600/200/300 mg for 96 weeks.
- EFV/TDF/FTC 600/200/300 mg Once Daily: During double-blind phase, participants received EFV/TDF/FTC 600/200/300 mg OD, with placebo to match DTG 50 mg and ABC/3TC 600/300 mg for 96 weeks.
Period: Double-blind Phase: 96 Weeks Duration
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Started | 414 | 419
Completed | 342 | 310
Not Completed | 72 | 109
Not completed — Adverse Event | 13 | 48
Not completed — Lack of Efficacy | 18 | 14
Not completed — Protocol Violation | 14 | 12
Not completed — Lost to Follow-up | 17 | 18
Not completed — Withdrawal by Subject | 9 | 15
Not completed — Physician Decision | 1 | 2
Period: Open-label Phase: 48 Weeks Duration
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Started | 341 | 309
Completed | 317 | 278
Not Completed | 24 | 31
Not completed — Adverse Event | 3 | 10
Not completed — Lack of Efficacy | 7 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 8 | 8
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily: During double-blind phase, participants received a dolutegravir (DTG) 50 milligram (mg) tablet along with an Abacavir/Lamivudine (ABC/3TC) 600/300 mg tablet once daily (OD) orally, with placebo to match Efavirenz/Tenofovir disoproxil fumarate/Emtricitabine (EFV/TDF/FTC) 600/200/300 mg for 96 weeks. Participants who completed double-blind phase continued to receive DTG 50 mg tablet along with ABC/3TC 600/300 mg tablet OD orally, for additional 48 weeks during open-label phase.
- EFV/TDF/FTC 600/200/300 mg Once Daily: During double-blind phase, participants received EFV/TDF/FTC 600/200/300 mg OD, with placebo to match DTG 50 mg and ABC/3TC 600/300 mg for 96 weeks. Participants who completed double-blind phase continued to receive EFV/TDF/FTC 600/200/300 mg OD for additional 48 weeks during open-label phase.
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily | Total
Number analyzed (Participants) | 414 | 419 | 833
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (10.74) | 36.4 (10.43) | 36.4 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 63 | 130
  Male | 347 | 356 | 703
Race/Ethnicity, Customized [Number; unit: participants]
  African American (Af Am)/African Heritage (Af Ht) | 98 | 99 | 197
  American Indian (AI) or Alaska Native (Nat) | 13 | 17 | 30
  Asian | 9 | 9 | 18
  White | 284 | 285 | 569
  Af Am/Af Ht & AI or Alaska Native | 0 | 1 | 1
  Af Am/Af Ht & Nat Hawaiian/other Pacific Islander | 0 | 1 | 1
  Af Am/Af Ht & White | 3 | 2 | 5
  American Indian or Alaska Native & White | 6 | 4 | 10
  Asian & White | 1 | 0 | 1
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Responding Based on Plasma HIV-1 RNA <50 c/mL at Week 48
Description: The percentage of participants with plasma HIV-1 RNA <50 c/mL at Week 48 was assessed. Plasma samples were collected for the quantitative assessment of HIV-1 RNA based on the Missing, Switch, or Discontinuation equals Failure (MSDF) algorithm,as codified by the Food and Drug Administration's Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigationl product prior to the visit window) as non-responders, as well as participants who switched their concomitant antiretroviral therapy (ART) in certain scenarios. Since changes in ART were not permitted in this protocol, all such participants who changed ART were to be considered non-responders. Otherwise, virologic success or failure was to be determined by the last available HIV-1 RNA assessment while the participant was on treatment within the visit of interest window.
Time Frame: Week 48
Population: Intent-to-Treat-Exposed (ITT-E) Population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Percentage of participants | 88 | 81
Statistical Analysis 1: Comparison: DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily vs EFV/TDF/FTC 600/200/300 mg Once Daily; Test type: Non-Inferiority or Equivalence — Non-inferiority could be concluded if the lower bound of a two-sided 95% confidence interval for the difference (DTG + ABC/3TC minus EFV/TDF/FTC) in percentages between the two treatment arms was > -10%; p = 0.003, Wilcoxon (Mann-Whitney) — P-value is for the test of superiority; Difference in percentage = 7.3, 95% CI 2-sided [2.3 to 12.2] — The estimated value reflects the percentage on DTG + ABC/3TC minus the percentage on EFV/TDF/FTC

2. Secondary Outcome: Time to Viral Suppression (<50 c/mL)
Description: Viral suppression is defined as the first viral load value<50 c/mL. The Kaplan-Meier method was used to estimate time to viral suppression, defined as the time from the first dose of study treatment until the first viral load value <50 c/mL was reached. Participants who withdrew for any reason without having suppressed prior to the analysis were censored.
Time Frame: From Baseline until Week 144) (average of 877.4 days for DTG; average of 788.8 study days for EFV/TDF/FTC)
Population: ITT-E Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Days | 28 [28.0 to 29.0] | 84 [83.0 to 84.0]

3. Secondary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus -1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) at Week 96 and Week 144
Description: The percentage of participants with plasma HIV-1 RNA <50 c/mL at Week 96 and Week 144 was assessed. Plasma samples were collected for the quantitative assessment of HIV-1 RNA based on the Missing, Switch, or Discontinuation equals Failure (MSDF) algorithm,as codified by the Food and Drug Administration's Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigationl product prior to the visit window) as non-responders, as well as participants who switched their concomitant antiretroviral therapy (ART) in certain scenarios. Since changes in ART were not permitted in this protocol, all such participants who changed ART were to be considered non-responders. Otherwise, virologic success or failure was to be determined by the last available HIV-1 RNA assessment while the participant was on treatment within the visit of interest window.
Time Frame: Week 96 and Week 144
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Percentage of participants
  Week 96 | 77 | 70
  Week 144 | 71 | 63
Statistical Analysis 1: Comparison: DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily vs EFV/TDF/FTC 600/200/300 mg Once Daily; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.016, Wilcoxon (Mann-Whitney) — P-value is for the test of superiority; Difference in percentage = 7.1, 95% CI 2-sided [1.2 to 13.1] — Week 96:The estimated value reflects the percentage on DTG + ABC/3TC minus the percentage on EFV/TDF/FTC
Statistical Analysis 2: Comparison: DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily vs EFV/TDF/FTC 600/200/300 mg Once Daily; Test type: Non-Inferiority or Equivalence — Non-inferiority could be concluded if the lower bound of a two-sided 95% confidence interval for the difference (DTG + ABC/3TC minus EFV/TDF/FTC) in percentages between the two treatment arms was >-10%; p = 0.010, Wilcoxon (Mann-Whitney) — P-value is for the test of superiority; Difference in percentage = 8.3, 95% CI 2-sided [1.9 to 14.6] — Week 144:Estimated value reflects the percentage on DTG + ABC/3TC minus the percentage on EFV/TDF/FTC

4. Secondary Outcome: Number of Participants With a Confirmed Plasma HIV-1 RNA Level >=1000 c/mL at or After Week 16 and Before Week 24, or a Confirmed Plasma HIV-1 RNA Level >=200 c/mL at or After Week 24
Description: Data are presented as Kaplan Meier estimates of virologic failure (VF), defined as a confirmed plasma HIV-1 RNA level >=1000 c/mL at or after Week 16 and before Week 24, or a confirmed plasma HIV-1 RNA level >=200 c/mL at or after Week 24. A plasma HIV-1 RNA value was considered to be confirmed failure if a consecutive measurement satisfied the same failure criterion. The number of participants who experienced autoimmune deficiency syndrome (AIDS) Clinical Trials Group (ACTG) VFs was measured. For participants who withdrew from the study/were not documented to have reached confirmed VF at the cut off date of the Week 48 analysis, time to VF was to be censored at the planned visit week of the last measured plasma HIV-1 RNA sample. Data for participants who missed three consecutive scheduled plasma HIV-1 RNA measurements were to be censored at the planned visit week of the last assessment prior to the 3 consecutive missed visits.
Time Frame: From Baseline until Week 144) (average of 877.4 days for DTG; average of 788.8 study days for EFV/TDF/FTC)
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Participants
  ACTG virologic failures | 11 (0.58) | 8 (0.52)
  Censored participants | 403 (0.70) | 411 (0.63)

5. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA at Weeks 2, 4, 8, 12, 16, 24, 32, 40,48, 60, 72, 84, 96, 108, 120, 132 and 144
Description: Blood samples were collected for the measurement of HIV-1 RNA in plasma. Changes from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants available at the indicated time points were assessed (represented by n=X, X in the category titles).
Time Frame: Baseline and at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
log10 copies/mL
  Week 2, n=387, 376 | -2.46 (0.49) | -1.96 (0.46)
  Week 4, n=404, 391 | -2.88 (0.58) | -2.25 (0.52)
  Week 8, n=395, 386 | -2.99 (0.64) | -2.60 (0.60)
  Week 12, n=394, 377 | -3.01 (0.70) | -2.85 (0.63)
  Week 16, n=386, 366 | -3.03 (0.66) | -2.98 (0.65)
  Week 24, n=389, 364 | -3.05 (0.69) | -3.01 (0.76)
  Week 32, n=380, 355 | -3.04 (0.70) | -3.05 (0.72)
  Week 40, n=370, 345 | -3.05 (0.68) | -3.04 (0.70)
  Week 48, n=370, 343 | -3.03 (0.69) | -3.04 (0.69)
  Week 60, n=360, 330 | -3.03 (0.67) | -3.05 (0.69)
  Week 72, n=354, 320 | -3.03 (0.70) | -3.06 (0.70)
  Week 84, n=353, 314 | -3.02 (0.70) | -3.07 (0.68)
  Week 96, n=345, 310 | -2.99 (0.73) | -3.06 (0.68)
  Week 108, n=340, 300 | -3.01 (0.71) | -3.08 (0.67)
  Week 120, n=333, 289 | -3.00 (0.77) | -3.07 (0.67)
  Week 132, n=323, 284 | -3.03 (0.68) | -3.06 (0.67)
  Week 144, n=313,269 | -3.02 (0.72) | -3.04 (0.69)

6. Secondary Outcome: Change From Baseline in CD4+ Cell Counts at Week 144
Description: Cluster of differentiation (CD4) lymphocyte cells (also called T-cells or T-helper cells) are the primary targets of HIV. The CD4 count and the CD4 percentage mark the degree of immunocompromise. The CD4 count is used to stage the patient's disease, determine the risk of opportunistic illnesses, assess prognosis, and guide decisions about when to start antiretroviral therapy. Change from Baseline was calculated as the Week 144 value minus the Baseline value. The least squares mean is the estimated mean change from Baseline in CD4+ cell counts at Week 144 calculated from a repeated measures model including the following covariates: treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, treatment*visit interaction, Baseline HIV-1 RNA*visit interaction, and Baseline CD4+ cell count*visit interaction. No assumptions were made about the correlations between a participant's readings of CD4+, i.e., the correlation matrix for within-participant errors is unstructured.
Time Frame: Baseline and Week 144
Population: ITT-E Population
Measure: Least Squares Mean (Standard Deviation); unit: cells per millimeters cubed (cells/mm^3)
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
cells per millimeters cubed (cells/mm^3) | 378.48 (10.99) | 331.57 (11.59)
Statistical Analysis 1: Comparison: DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily vs EFV/TDF/FTC 600/200/300 mg Once Daily; Test type: Non-Inferiority or Equivalence — Adjusted mean is the estimated mean change from baseline (BL) in CD4 + Cell Count at Week 144 in each arm calculated from a repeated measures model including the following covariates: treatment, visit, BL plasma HIV-1 RNA, BL CD4 cell count, treatment*visit interaction, BL HIV-1 RNA*visit interaction and BL CD4 cell count*visit interaction. No assumptions were made about the correlations between a par.'s readings of CD4 i.e. the correlation matrix for within-subject errors is unstructured; p = 0.003, Repeated Measure Mixed Model — P-value is for the test of superiority

7. Secondary Outcome: Change From Baseline in CD4+ Cell Counts at Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144
Description: CD4 lymphocyte cells (also called T-cells or T-helper cells) are the primary targets of HIV. The CD4 count and the CD4 percentage mark the degree of immunocompromise. The CD4 count is used to stage the patient's disease, determine the risk of opportunistic illnesses, assess prognosis, and guide decisions about when to start antiretroviral therapy. Change from Baseline was calculated as the value at Indicated visit minus the Baseline value. Only those participants available at the indicated time points were assessed (represented by n=X, X in the category titles).
Time Frame: Baseline and Week 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: cells per millimeters cubed (cells/mm^3)
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
cells per millimeters cubed (cells/mm^3)
  Week 4, n=404,390 | 117.6 (114.51) | 80.9 (112.43)
  Week 8, n=396,382 | 164.6 (129.98) | 124.4 (124.50)
  Week 12, n=394,378 | 187.5 (157.46) | 153.0 (131.91)
  Week 16, n=386,366 | 214.7 (173.35) | 174.1 (132.02)
  Week 24, n=388,361 | 216.9 (162.89) | 177.8 (147.72)
  Week 32, n=380,353 | 250.5 (172.06) | 208.1 (152.13)
  Week 40, n=364,347 | 265.5 (187.81) | 216.2 (158.49)
  Week 48, n=368,344 | 267.5 (192.30) | 209.5 (164.37)
  Week 60, n=359,330 | 271.3 (188.05) | 235.3 (171.98)
  Week 72, n=354,319 | 306.1 (202.02) | 269.6 (180.04)
  Week 84, n=352,314 | 315.2 (197.92) | 272.1 (172.28)
  Week 96, n=343,309 | 322.6 (205.35) | 286.0 (195.70)
  Week 108, n=339,300 | 349.3 (218.76) | 298.9 (188.41)
  Week 120, n=332,287 | 347.0 (234.96) | 311.0 (198.79)
  Week 132, n=323,283 | 377.9 (205.78) | 327.2 (175.31)
  Week 144, n=313,270 | 379.5 (221.17) | 333.3 (189.25)

8. Secondary Outcome: Number of Participants With the Indicated Post-baseline HIV-associated Conditions and Progression, Excluding Recurrences at Week 144
Description: Clinical disease progression (CDP) was assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the AIDS surveillance case definition. Indicators of CDP were defined as: CDC CAT A at Baseline (BS) to a CDC CAT C event (EV); CDC CAT B at BS to a CDC CAT C EV; CDC CAT C at BS to a new CDC CAT C EV; or CDC CAT A, B, or C at BS to death.
Time Frame: From Baseline until Week 144
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Participants
  Week 144, Any category condition | 17 | 24
  Week 144, Any Category B condition | 12 | 17
  Week 144, Any Category C condition | 5 | 6
  Week 144, Any death | 0 | 2
  Week 144, Progression from CAT A to CAT C | 4 | 4
  Week 144, Progression from CAT C to new CAT C | 1 | 2
  Week 144, Progression from CAT A, B, or C to death | 0 | 2

9. Secondary Outcome: Number of Participants With the Indicated Grade 1 to 4 Clinical and Hematology Toxicities at Week144
Description: All Grade 1 to 4 post-Baseline-emergent chemistry toxicities included alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), asparate aminotransferase (AST), carbon dioxide (CO2) content/bicarbonate, cholesterol, creatine kinase (CK), creatinine, hyperglycemia, hyperkalemia, hypernatremia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) cholesterol calculation, lipase, phosphorus inorganic, total bilirubin, and triglycerides. All Grade 1 to 4 post-Baseline-emergent hematology toxities included hemoglobin, platelet count, total neutrophils, and white blood cell count. The Division of AIDS (DAIDS) defined toxicity grades as follows: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening; Grade 5, death.
Time Frame: From Baseline until Week 144
Population: Safety Population: all participants who received at least one dose of investigational product
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 414 | 419
Participants
  Week 144, ALT | 62 (0.3849) | 81 (0.3854)
  Week 144, Albumin | 0 | 1
  Week 144, ALP | 17 | 53
  Week 144, AST | 77 | 85
  Week 144, CO2 content/bicarbonate | 135 | 134
  Week 144, Cholesterol | 156 | 140
  Week 144, CK | 91 | 79
  Week 144, Creatinine | 17 | 6
  Week 144, Hyperglycaemia | 121 | 105
  Week 144, Hyperkalemia | 4 | 12
  Week 144, Hypernatremia | 11 | 9
  Week 144, Hypoglycaemia | 24 | 21
  Week 144, Hypokalemia | 38 | 21
  Week 144, Hyponatremia | 63 | 86
  Week 144, LDL cholesterol calculation | 124 | 111
  Week 144, Lipase | 111 | 110
  Week 144, Phosphorus, inorganic | 109 | 134
  Week 144, Total bilirubin | 22 | 4
  Week 144, Triglycerides | 11 | 11
  Week 144, Hemoglobin | 7 | 11
  Week 144, Platelet count | 20 | 19
  Week 144, Total neutrophils | 70 | 80
  Week 144, White Blood Cell count | 9 | 18

10. Secondary Outcome: Number of Participants With the Indicated Genotypic Resistance With Virological Failure (VF) Through 144
Description: Whole blood samples were collected from participants to provide plasma for storage samples for potential viral genotypic and phenotypic analyses. Participants with confirmed virological failure (confirmed HIV-1 RNA >=50 copies/mL throughout the study and/or confirmed HIV-1 RNA >=200 copies/mL at Week 144) had plasma samples tested for HIV-1 RT genotype and HIV-1 integrase genotype from Baseline samples and from samples collected at the time of virological failure. Genotype testing was conducted at Day 1 and at the time of suspected protocol-defined virological failure (PDVF). A genotyping assessment was made of change across all amino acids within the integrase (IN)-encoding region, with particular attention paid to specific amino acid changes associated with the development of resistance to RAL, ELV, or DTG.
Time Frame: Through Week 144
Population: PDVF Genotypic Population: all participants in the ITT-E Population with available on-treatment genotypic resistance data at the time of PDVF
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 26 | 16
Participants
  Week 144, RT mutation K65K/R | 0 | 1
  Week 144, RT mutation K101E | 0 | 1
  Week 144, RT mutation K103K/N | 0 | 2
  Week 144, RT mutation K103N | 0 | 2
  Week 144, RT mutation G190G/A | 0 | 2

11. Secondary Outcome: Change From Baseline in the Symptom Bother Score (SBS) at Week 4 Through Week 48
Description: The Symptom Distress Module (SDM) is a 20-item, self-reported questionnaire measuring the presence/perceived distress linked to symptoms associated with HIV/its treatments. Developed with support from the AIDS Clinical Trials Group of the U.S. National Institute of Allergy and Infectious Diseases, it has demonstrated construct validity and has shown strong associations with physical/mental health summary scores and with disease severity. The SDM consists of 2 main scores: symptom count and the SBS, ranging from 0 (best) to 80 (worst) and based on the degree of bother that each symptom present posed. The SBS was calculated by adding the 20 individual bother item scores, which were calculated as: 0, "I do not have this symptom"; 1, "It doesn't bother me"; 2, "It bothers me a little"; 3, "It bothers me"; 4, "It bothers me a lot." Estimates are calculated from an analysis of covariance (ANCOVA) model adjusting for age, sex, race, Baseline (BL) viral load, BL CD4+ cell count, and BL SBS.
Time Frame: Baseline and Week 4 through 48
Population: ITT-E Population. Participants with missing bother item scores at Week 4 had their last observation carried forward (LOCF). Only those participants contributing to the model (i.e., without missing response variables after LOCF or covariates) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Number analyzed (Participants) | 394 | 393
Scores on a scale | -1.818 (0.3849) | -1.246 (0.3854)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to Week 144 (average of 877.4 study days for DTG; average of 788.8 study days for EFV/TDF/FTC).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily | EFV/TDF/FTC 600/200/300 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 65/414 | 60/419
Other Adverse Events (participants affected / at risk) | 332/414 | 358/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily (N=414) | EFV/TDF/FTC 600/200/300 mg Once Daily (N=419)
Pneumonia (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 3
Syphilis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 4 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 3
Systemic candida (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 2
Suicide attempt (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 3
Homicidal ideation (Psychiatric disorders) | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2
AIDS dementia complex (Infections and infestations) | 0 | 1
Cellulitis pharyngeal (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Human herpesvirus 6 infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Shared psychotic disorder (Psychiatric disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 3
Coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Adverse drug reaction (General disorders) | 1 | 0
Systemic inflammatory response sydrome (General disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg Plus ABC/3TC 600/300 mg Once Daily (N=414) | EFV/TDF/FTC 600/200/300 mg Once Daily (N=419)
Dizziness (Nervous system disorders) | 43 | 154
Headache (Nervous system disorders) | 67 | 64
Somnolence (Nervous system disorders) | 10 | 24
Insomnia (Psychiatric disorders) | 74 | 52
Abnormal dreams (Psychiatric disorders) | 32 | 74
Depression (Psychiatric disorders) | 34 | 38
Anxiety (Psychiatric disorders) | 33 | 35
Diarrhoea (Gastrointestinal disorders) | 94 | 89
Nausea (Gastrointestinal disorders) | 70 | 63
Nasopharyngitis (Infections and infestations) | 86 | 81
Upper respiratory tract infection (Infections and infestations) | 69 | 58
Fatigue (General disorders) | 67 | 56
Pyrexia (General disorders) | 27 | 30
Rash (Skin and subcutaneous tissue disorders) | 22 | 63
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 40
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 25
Nightmare (Psychiatric disorders) | 11 | 21
Vomiting (Gastrointestinal disorders) | 28 | 27
Bronchitis (Infections and infestations) | 33 | 33
Syphilis (Infections and infestations) | 26 | 31
Sinusitis (Infections and infestations) | 29 | 18
Influenza (Infections and infestations) | 31 | 14
Gastroenteritis (Infections and infestations) | 26 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 | 19
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.